CLINICAL TRIAL: NCT06261021
Title: A Phase 2, Single-Blind, Intraindividual Study to Evaluate the Efficacy of Ruxolitinib 1.5% Cream in Adult Subjects with Discoid Lupus Erythematosus
Brief Title: Study to Evaluate the Efficacy of Ruxolitinib 1.5% Cream in Adult Subjects with Discoid Lupus Erythematosus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INNO-6051
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Discoid Lupus Erythematosus
Keywords: discoid lupus erythematosus; opzelura; ruxolitinib cream
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — ruxolitinib; Salicylic Acid

STUDY DESIGN:
Intervention Model Description: Intra-individual
Who Masked: Outcomes Assessor
Masking Description: This study will be single-blinded. Only the efficacy assessor will be blinded in this study (for subjects with randomized areas). The assessor will only assess efficacy and will not have any other interactions with the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ruxolitinib 1.5% cream (Sequence 1) (Experimental): ruxolitinib 1.5% cream without occlusion for Area 1 and ruxolitinib 1.5% cream under occlusion at night for Area 2
  Interventions: Drug: Ruxolitinib 1.5% cream; Procedure: Application without occlusion in Area 1; Procedure: Application under occlusion at night in Area 2
- ruxolitinib 1.5% cream ( Sequence 2) (Experimental): ruxolitinib 1.5% cream under occlusion at night for Area 1 and ruxolitinib 1.5% cream without occlusion for Area 2
  Interventions: Drug: Ruxolitinib 1.5% cream; Procedure: Application under occlusion at night in Area 1; Procedure: Application without occlusion in Area 2

INTERVENTIONS:
Drug: Ruxolitinib 1.5% cream — Topical application of Ruxolitinib 1.5% cream
Procedure: Application without occlusion in Area 1 — Apply Ruxolitinib 1.5% cream on the discoid lupus erythematosus lesion without occlusion on Area 1.
  Arms: ruxolitinib 1.5% cream (Sequence 1)
Procedure: Application under occlusion at night in Area 2 — Apply Ruxolitinib 1.5% cream on the discoid lupus erythematosus lesion under occlusion at night on Area 2.
  Arms: ruxolitinib 1.5% cream (Sequence 1)
Procedure: Application under occlusion at night in Area 1 — Apply Ruxolitinib 1.5% cream on the discoid lupus erythematosus lesion under occlusion at night on Area 1.
  Arms: ruxolitinib 1.5% cream ( Sequence 2)
Procedure: Application without occlusion in Area 2 — Apply Ruxolitinib 1.5% cream on the discoid lupus erythematosus lesion without occlusion on Area 2.
  Arms: ruxolitinib 1.5% cream ( Sequence 2)

SUMMARY:
This study is a single-blind, intraindividual study to evaluate the efficacy of ruxolitinib 1.5 % cream in adult subjects with discoid lupus erythematosus.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the efficacy, safety and tolerability of ruxolitinib 1.5 % cream in adult subjects with discoid lupus erythematosus.

Approximately 20 subjects with discoid lupus erythematosus will apply ruxolitinib 1.5% cream, twice daily on active lesions identified at Day 1 and any new lesions that appear, for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 years of age or older at the time of consent.
* Confirmed DLE diagnosis.
* Subject has moderate to severe DLE, as defined by an overall CLA IGA score of 3 (moderate) or 4 (severe) at screening and Day 1.
* Female subject of childbearing potential must have a negative urine pregnancy test at screening and negative urine pregnancy test at Day 1.
* Subject has no known history of latent or active tuberculosis (TB) infection.
* Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
* Subjects must be willing to comply with all study procedures and must be available for the duration of the study.

Exclusion Criteria:

* Female subject who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
* Subject has a history of skin disease or presence of skin condition that would interfere with the study assessments.
* Subject has unstable or fluctuating use of nicotine-containing products within 4 weeks prior to screening.
* Subject is known to have immune deficiency or is immunocompromised.
* Subject is ≥ 50 years old AND has a history of heart attack, other clinically significant heart problems, stroke, or blood clots.
* Subject has a known history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus [HIV]).
* Subject is known to have hepatitis B or hepatitis C viral infection.
* Subject has used any topical medicated treatment that could affect DLE within 2 weeks prior to Day 1, including, but not limited to, topical corticosteroids, retinoids, calcineurin inhibitors, antimicrobials, and medical devices.
* Subject has received any marketed or investigational biological agent within 12 weeks or 5 half lives (whichever is longer) prior to Day 1, including but not limited to ustekinumab and rituximab.
* Subject is currently receiving a nonbiological investigational product or device or has received one within 4 weeks prior to Day 1.
* Subject has a known or suspected allergy to ruxolitinib.
* Subject has used ruxolitinib cream (OpzeluraTM).
* Subject has used JAK inhibitors for conditions other than DLE or other forms of lupus within 4 weeks prior to Day 1.
* Subject has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in target lesion CLASI-A score | Week 24
  The CLASI-A (Cutaneous Lupus Area and Severity Index - Activity) quantifies disease activity based on scoring of erythema, scale/hypertrophy, mucous membrane involvement, acute hair loss, and non scarring alopecia.
  Change from baseline in target lesion CLASI-A score at Week 24 for the target DLE lesion treated with occlusion The CLASI-A score ranges from 0 to 70, with higher scores indicating more severe skin disease.

SECONDARY OUTCOMES:
Change from baseline in target lesion CLASI-A score | Week 12, Week 24
  The CLASI-A (Cutaneous Lupus Area and Severity Index - Activity) quantifies disease activity based on scoring of erythema, scale/hypertrophy, mucous membrane involvement, acute hair loss, and non scarring alopecia.
  Change from baseline in target lesion CLASI-A score at Week 24 for the target DLE lesion treated without occlusion.
  The CLASI-A score ranges from 0 to 70, with higher scores indicating more severe skin disease.
Proportion of subjects with an erythema score of 0 (absent) | Week 24
  Proportion of subjects with an erythema score of 0 (absent) in 50% of all DLE lesions. Erythema will be assessed for each DLE lesion identified on Day 1 using the erythema component of the CLASI-A scale. The severity of erythema is scored on a 4-point scale ranging from 0 (absent) to 3.
Change from baseline in target lesion SADDLE-A | Week 12, Week 24
  Change from baseline in target lesion SADDLE-A at Week 24 for the target DLE lesion treated with and without occlusion.
  Change from baseline in target lesion SADDLE-A score at Week 12 for the untreated target DLE lesion and the target DLE lesion treated with and without occlusion
Proportion of subjects with a target lesion CLA-IGA score of 0 (clear) or 1 (almost clear) | Week 24
  Proportion of subjects with a CLA-IGA score of 0 (clear) or 1 (almost clear) for all DLE lesions. The CLA-IGA is a 5 point scale that evaluates the severity of signs of the overall disease activity based on erythema, scale, edema/ infiltration, follicular involvement, and secondary changes.

OTHER OUTCOMES:
Dermatology Life Quality Index (DLQI) | Weeks 12 and 24
  Change from baseline in DLQI. Quality of life will be evaluated using Dermatology Life Quality Index (DLQI). It is a simple 10-question validated questionnaire that has been used in more than 40 different skin conditions.The DLQI is the most frequently used instrument in studies of randomized controlled trials in dermatology.
Cutaneous Lupus Erythematosus Quality of Life (CLEQol) | Weeks 12 and 24
  Change from baseline in CLEQoL total score.Quality of life will be evaluated using the Cutaneous Lupus Erythematosus Quality of Life (CLEQoL).The CLEQoL asks subjects to assess how often (never, rarely, sometimes, often, all the time) they experienced a given effect. Scores of 0 (never), 25 (rarely), 50 (sometimes), 75 (often), or 100 (all the time) are assigned to each question. The scores are averaged per domain from the scale of 0-100, with higher numbers indicating worse quality of life.
Numeric Rating Scale(NRS) | Weeks 12 and 24
  Change from baseline in target lesion pruritus NRS scores.Pruritus numeric rating scale (NRS) will also be evaluated as an efficacy assessment for each of the 2 (or 3, as applicable) target lesions.This will be evaluated by asking subjects to assign a numerical score representing worst itch intensity over the last 24 hours of each target lesion on a scale from 0 to 10, with 0 indicating no itch and 10 indicating the worst imaginable itch.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.
Locations (2):
- Canada (2):
  - INNO-6051 Site 03, Fredericton, New Brunswick
  - Innovaderm Research Inc., Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No